CLINICAL TRIAL: NCT02924220
Title: Genetic Susceptibility and Biomarkers in Listeriosis (MONALISA-GENBIO)
Brief Title: Genetic Susceptibility and Biomarkers in Listeriosis
Acronym: MONALISAGENBIO
Status: Completed | Type: Observational
Sponsor: Institut Pasteur (Industry)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-038; ID-RCB number : 2016-A00650-51 (Other: French national registration number of the study)
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Listeriosis
MeSH Terms: conditions — Listeriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Biological samples (serum, plasma, mononuclear cells and DNA) previously collected from cases patients and control patients included in the MONALISA cohort.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case patients: Patients with culture-proven listeriosis. Case patients are classified in 3 groups :
  * Septicemic infections: isolation of Lm in blood cultures.
  * CNS infections: isolation of Lm in cerebrospinal fluid, or brain stereotaxic biopsy, or by isolation of Lm in the blood with concomitant meningitis, or radiological encephalitis, rhombencephalitis, brain abscess or meningitis.
  * MF infections: defined by isolation of Lm in any maternal/fetal/neonatal bacteriological sample.
  All patients have given their written consent to participate in the MONALISA cohort and for the collection of a blood sample including DNA samples for DNA analyses will be included in the MONALISA GENBIO study.
- Control patients: Patients without listeriosis but compatible clinical presentation. Control patients are divided in 3 groups.
  * Septicemic controls: febrile patient with same co-morbidities as septicemic cases.
  * CNS controls: patient with any neurological symptom leading to the empiric prescription of amoxicillin at meningeal dosage because of listeriosis presumption.
  * MF controls: febrile pregnant patient without obvious focal infection.
  All patients have given their written consent to participate in the MONALISA cohort and for the collection of a blood sample including DNA samples for DNA analyses will be included in the MONALISA GENBIO study.

SUMMARY:
Listeriosis is a rare, severe foodborne infection caused by the bacterium Listeria monocytogenes (Lm). It manifests as septicemia, central nervous system (CNS) infection and maternal-fetal (MF) infection. Its associated overall mortality is very high, above of 30%. A better knowledge on the factors involved in its occurrence and in clinical manifestations is therefore needed to improve outcome.

A number of frequent acquired risk factors for listeriosis have been identified, such as pregnancy, diabetes, cancer, HIV infection, and immunosuppressive therapies. However, no genetic study on host susceptibility to listeriosis in humans has been performed so far, in the absence of prospective collection of patients' samples. Also, listeriosis diagnosis is based on Lm culture from clinical samples. This method lacks sensitivity, and the contribution of biomarkers to listeriosis diagnosis and prognosis has not been evaluated.

The Multicentric Observational NAtional Analysis of Listeriosis and Listeria (MONALISA), is the first national case-control prospective study on listeriosis. It is implemented since 2009 and enrolls all culture-proven cases declared to the NRCL: and collects for each patient clinical and biological data and biological samples. Controls with comparable background and presentation are also included. 818 cases have been included (427 S, 252 CNS and 107 MN) over 3.5 years, along with 456 controls.

The aim of the study is to identify human genetic susceptibility factors to listeriosis, biomarkers to improve its diagnosis and prognosis (survival or death), and thereby help improve management of patients with listeriosis.

Samples from the completed cohort will be analyzed : SNPs genotyping and exam sequencing; biomarkers a identification in serum and plasma of patients and controls by simultaneous multi-analyte and metabolomic profiling.

DETAILED DESCRIPTION:
Context :

Listeriosis is a rare, severe foodborne infection caused by the bacterium Listeria monocytogenes (Lm). It manifests as septicemia, central nervous system (CNS) infection and maternal-fetal (MF) infection. Its associated overall mortality is very high, above of 30%. A better knowledge on the factors involved in its occurrence and in clinical manifestations is therefore needed to improve outcome. Surveillance of human listeriosis in France relies on the mandatory reporting of cases and the submission of the corresponding Lm strains to the National Reference Centre for Listeria (NRCL).

A number of acquired risk factors for listeriosis have been identified, such as pregnancy, age, cirrhosis, renal insufficiency, diabetes, cancer, HIV infection, transplantation and immunosuppressive therapies. If listeriosis is rare, the exposure to Lm is universal. The high prevalence of known risk factors in the general population and the low occurrence of the disease suggest that unknown parameters, such as host genetic factors, contribute to the susceptibility to listeriosis. This is supported by animal studies, which have shown that genes involved in innate and cell-based immunity are critical to control listeriosis. However, no genetic study on host susceptibility to listeriosis in humans has been performed so far, in the absence of prospective collection of patients' samples.

Listeriosis diagnosis is based on Lm culture from clinical samples. This specific method lacks sensitivity, and the usefulness of PCR or serological assays have not been assessed in prospective case-control studies. Biomarkers are useful tools to diagnose infections and assess their severity, but their contribution to listeriosis diagnosis and prognosis has not been evaluated.

The Multicentric Observational NAtional Analysis of Listeriosis and Listeria (MONALISA), a national case-control prospective study on listeriosis, was launched in 2009. It enrolls all culture-proven cases declared to the NRCL: clinical and biological data and biological samples (plasma, serum, PBMC) are collected at inclusion for each patient. Controls with comparable background and presentation are also included. 818 cases have been included (427 S, 252 CNS and 107 MN) over 3.5 years, along with 456 controls.

Hypothesis :

* host genetic variation plays an important role in determining susceptibility to listeriosis and its clinical manifestations. Common host genetic variation in the human population may play a role in susceptibility in association with known acquired risk factors. Rare variants may also explain severe manifestations of listeriosis, such as death, severe persistent neurological impairment and fetal loss, in the absence of risk factors.
* biomarker patterns can assess and predict infection and infection severity. Immune responses may be tracked as a biological signature of invasive listeriosis
* biomarkers patterns could hopefully correlate with genotypic characterization as a phenotypic reflection of a genetically inadequate / missing link hampering the proper coordination of the immune response to Lm.

Methods :

* SNP arrays genotyping of the whole cohort
* Whole-exome sequencing of the whole cohort to identify rare variants
* Biomarkers identification in serum and plasma of patients and controls by simultaneous multi-analyte and metabolomic profiling:

The cohort is already constituted.

Expected results :

Better understanding of major biomedical aspects of listeriosis, namely host genetic susceptibility factors and diagnostic/prognostic biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* All patients have given their written consent to participate in the MONALISA cohort and for the collection of a blood sample including DNA samples for DNA analyses.

Exclusion Criteria:

* Patients included in the MONALISA cohort without biological sample available.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients already recruited in the MONALISA study will be included. The MONALISA study is the first prospective case-control study focused on invasive listeriosis. Cases are patients with culture-proven listeriosis. Controls are patients without listeriosis but compatible clinical presentation.
Sampling Method: Non-Probability Sample
Enrollment: 1080 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Characterisation of genetic susceptibility markers for infection as a whole and for each form and/or for the severity of infection | 3 years
  Characterisation of genetic susceptibility markers for infection as a whole and for each form and/or for the severity of infection by whole exome sequencing and whole genome genotyping for all MONALISA cases and controls

SECONDARY OUTCOMES:
Biomarkers identification in serum and plasma of patients and controls | 3 years
  Biomarkers identification in serum and plasma of patients and controls by simultaneous multi-analyte and metabolomic profiling:
  -Characterisation of a biological signature of listeriosis as a whole and for each form of infection.
Biomarkers identification in serum and plasma of patients and controls | 3 years
  Biomarkers identification in serum and plasma of patients and controls by simultaneous multi-analyte and metabolomic profiling:
  -Characterisation of the severity of infection (prognosis): death, fetal loss, neurological persisting impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Lecuit, Study Director — Institut Pasteur
Locations (1):
- Institut Pasteur, Unité de Biologie des Infections, Paris, France

IPD SHARING:
Plan to Share IPD: No